CLINICAL TRIAL: NCT02337023
Title: Brain Scintigraphy in Normal Versus Kleine-Levin Syndrome Subjects
Acronym: SCINTIK
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P101002
Record Dates: First submitted 2014-12-05; First posted 2015-01-13 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Subjects; Kleine-Levin Syndrome
Keywords: Brain scintigraphy
MeSH Terms: conditions — Kleine-Levin Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy subjects
  Interventions: Radiation: Brain scintigraphy with injection of Neurolite® (ECD)
- patients with Kleine-Levin Syndrome
  Interventions: Radiation: Brain scintigraphy with injection of Neurolite® (ECD)

INTERVENTIONS:
Radiation: Brain scintigraphy with injection of Neurolite® (ECD) — Brain scintigraphy with injection of Neurolite® (ECD) 1 injection

SUMMARY:
The investigators perform neuropsychological tests and brain scintigraphy in 30 healthy subjects.

These results will be compared with data obtained out of episode in patients with Kleine-Levin syndrome (KLS).

The investigators want to determine if brain functional imaging and cognitive abnormalities persist during asymptomatic period in a large series of patients with KLS, and to find predictors of these abnormalities.

DETAILED DESCRIPTION:
3 steps in the protocol :

* Brain ECD-SPECT (marking brain perfusion in relation to brain active/hypoactive area) superimposed on a template T1-weighted brain MRI.
* Extensive cognitive tests of executive functions, verbal memory and fluency , visuospatial ability and memory, reasoning abilities: spontaneous memory complaint, Stroop Color Word Test, Trail Making Test A and B, Direct and Reverse Digit Span Test, Letter and Semantic Fluency Test, Free and Cued Selective Reminding Test, Rey-Osterrieth Complex Figure, Mini-Mental test, Progressive matrice of Raven (PM-38)
* KLS-inventory and face to face interview of patients and parents by neurologist for patients. Modified KLS-inventory for healthy subjects.

Main outcome : Number of patients with persisting hypoperfused brain area (compared to controls), location of these area, number of patients with at least -1SD in one cognitive domain Correlation between KLS severity (disease course, number of episode, mean duration of episodes, time incapacitated, number of symptoms) and brain perfusion and cognitive abnormalities

ELIGIBILITY:
Inclusion criteria :

* Subjects males and females with more than 18 y.o, age and sex-matched with patients with Kleine-Levin Syndrome
* with the same educational level and dominant hand than patients with Kleine-Levin Syndrome
* without any brain disease or sleep disease (Epworth score < 11/24) known.
* with social security
* french language
* for women : nonpregnant taking effective contraception

Exclusion criteria :

* Minor subjects
* adults under protection
* subjects with neurologic, psychiatric, somatic or sleep diseases and/or receiving a psychotropic medication interfering with the results.
* subjects with history of seizures or loss of consciousness
* subjects with excessive alcohol consumption (more than 3 doses /day)
* subjects without any social security
* subjects non fluent in french
* for women : no effective contraception or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Brain perfusion. | day 0
  Brain perfusion measured by scintigraphy with injection of Neurolite® (ECD) with a voxel by voxel approach

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ARNULF, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière, Paris, France